CLINICAL TRIAL: NCT03505307
Title: Lynparza Tablets 100mg, 150mg Clinical Experience Investigation (All Case Investigation) in Patients With Platinum-sensitive Relapsed Ovarian Cancer
Brief Title: Lynparza Ovarian Cancer Clinical Experience Investigation (All Case Investigation)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D0816C00019
Record Dates: First submitted 2018-04-10; First posted 2018-04-23 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
[Objectives] Objectives include following to capture safety and efficacy of LYNPARZA in actual clinical use.

1. ADR development in actual clinical use
2. Factors which may affect safety and efficacy
3. ADRs not expected from "Precautions for Use"

DETAILED DESCRIPTION:
The objective of the Clinical Experience Investigation (CEI) is to collect following data to characterise safety and efficacy of LYMPARZA Tablets 100mg and 150mg (LYMPARZA) in usual post-marketing use.

1. Development of adverse drug reactions (ADRs)
2. Factors which may affect safety and efficacy of LYMPARZA
3. Development of adverse drug reactions (ADRs) unexpected from "Precautions for Use" of the LYMPARZA JPI

ELIGIBILITY:
Inclusion Criteria:

* Maintenance treatment for patients with recurrent ovarian cancer, who are sensitive to platinum based chemotherapy

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with LYNPARZA for ovarian cancer which is the indication of the drug
Sampling Method: Non-Probability Sample
Enrollment: 846 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence of ADRs regarding Bone marrow depression, ILD, new primary malignancies, Embryo-foetal toxicity and exposure in patient with renal impairment | from baseline to 1 year
  To be calculated incidence of ADRs related to LYMPARZA during the observation period regarding Bone marrow depression, ILD, new primary malignancies, Embryo-foetal toxicity and exposure in patient with renal impairment
Factors which may impact incidence of ADRs related to LYMPARZA during the observation period, analysed by patient demographic characteristics | from baseline to 1 year
  Factors which may impact incidence of ADRs, analysed by patient demographic characteristic(past medical history, and concomitant disease etc)
Incidence of ADRs not expected from "Precautions for Use" of LYNPARZA JPI | from baseline to 1 year
  To be calculated incidence of ADRs related to LYMPARZA during the observation period not expected from "Precautions for Use" of LYNPARZA JPI

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00019&attachmentIdentifier=a365b2c5-bdad-46f6-aa6b-29f7046b1c7c&fileName=D0816C00019_CSR_Synopsis.pdf&versionIdentifier=
- See also: redacted protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00019&attachmentIdentifier=d760e7c1-913b-4778-9b10-10b914079225&fileName=D0816C00019_Protocol_redacted.pdf&versionIdentifier=